CLINICAL TRIAL: NCT05617092
Title: The Effect of a Postpartum Training Program on Women Who Have Suffered a Levator Ani Injury. A Pilot Randomized Controlled Trial Study
Brief Title: The Effect of a Postpartum Training Program on Women Who Have Suffered a Levator Ani Injury.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Rocio Montejo Rodriguez, PhD, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 278806
Record Dates: First submitted 2022-11-01; First posted 2022-11-15 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Pelvic Floor Disorders; Pelvic Floor; Perineal Rupture, Obstetric; Physiotherapy
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): intervention group will receive a physiotherapy individualized treatment
  Interventions: Other: Physiotherapy treatment
- Control Group (No Intervention): No intervention in women with injury in the levator ani
- Healthy controls (No Intervention): A group of women without injury that will be invited to filling in the questionnaires that will be carried out in the study three, six months and one year postpartum.

INTERVENTIONS:
Other: Physiotherapy treatment — physiotherapy individualized treatment according to the needs of the patient and clinical findings and symptoms
  Arms: Intervention group

SUMMARY:
The goal of this pilot randomized pilot controlled trial (RTC)is to collect acceptability and feasibility outcomes of a physiotherapy individualized program in women with levator injury that is intended to be used in a larger scale multicenter randomized controlled trial (RTC) in the future. The main questions it aims to answer are if a physiotherapy program in women with a levator injury:

1. Can improve the pelvic floor morphometry (PFM).
2. Can improve urogynecological symptoms
3. The effect of a physiotherapy program in the sexual function
4. The effect of a physiotherapy program in the patient's fear avoidance beliefs about physical activity and work Type of study: randomized pilot controlled trial (RTC) The design of this trial will be a pilot randomized controlled trial with 3 arms. Participants will be randomized in 2 arm of women with levator ani injury to either physiotherapy or standard care and an arm of woman without levator injury Researchers will compare the 3 groups to see if a physiotherapy program have benefits in morphometry of the pelvic floor, urogynecological symptoms, sexual function and to avoid fear avoidance beliefs about physical activity and work.

DETAILED DESCRIPTION:
The levator ani is a broad, thin muscle group, situated on either side of the pelvis. It supports the viscera in the pelvic cavity, and surrounds the various structures that pass through it. The levator ani muscles are of central importance in pelvic organ support and the maintenance of urinary and fecal continence. Vaginal delivery was associated with a higher number of pelvic floors injury at different levels (10% to 30% of women with vaginal deliveries). One of these specific types of pelvic floor injury include levator avulsion muscle (LAM) and levator ballooning. International clinical guidelines in agreement with meta-analysis recommend pelvic floor muscle (PFM) physiotherapy as a first line treatment for symptoms related to postpartum injuries. However, it is unclear whether women with levator ani injury lesions could respond to physiotherapy. There have been no randomized studies on this matter and the pilot studies have focused on anatomy rather than symptoms.

Trial Design A randomized pilot-controlled trial is designed to collect acceptability and feasibility outcomes of a physiotherapy individualized program in women with levator ani injury that is intended to be used in a larger scale multicenter randomized controlled trial in the future.

Methods The design of this trial will be a pilot randomized controlled trial with 3 arms:2 randomized arm of women with levator ani injury to either physiotherapy or standard care and an arm of woman without levator injury Participants Assessed for eligibility will be primiparous with a simplex vaginal delivery, aged ≥18 years, that understands the Swedish language, who approve vaginal examinations and with known risk factors for avulsion (instrumental delivery, maternal age >35 years, prolonged or precipitous second stage, and fetal occipito-posterior position).

10-12 weeks after the delivery a clinical 3 D ultrasound of pelvic floor will be perform.

Women with an injury in the levator ani will be randomized into two groups, one for intervention and the other for control.

Interventions The intervention group will receive a physiotherapy individualized treatment according to the needs of the patient and clinical findings and symptoms with the information provided by the employed questionnaires and clinic exploration.

Physiotherapy treatment will start from 3 months postpartum to about 1 year after The control group will receive general information according to the postpartum care guidelines of the region ( Västrä Gotaland Regionen).

Objective

The main objectives of this pilot study will be to evaluate the effect of a physiotherapy program in women with a levator ani injury:

1. To demonstrate the feasibility of conducting a trial to evaluate the intervention, including the feasibility and acceptability of randomising the intervention and the feasibility of outcome measure collection.
2. To improve the pelvic floor muscle morphometry.
3. To improve the urogynecological symptoms.
4. To improve the sexual function.
5. To improve the patient's fear avoidance beliefs about physical activity. Outcome Morphometrics variables as Pelvic Organ Prolapse Quantification Examination (POP-Q) Modified Oxford Grading System and Ultrasound variables: External an external sphincter, Levator hiatus area at rest (cm2),during Valsalva (cm2) and at maximum contraction (cm2) LAM area (cm2), Right and left puborectal muscle thickness (mm) will be collect.

The followed questionnaires will be use: Pelvic Floor Impact Questionnaire (PFIQ-7), Pelvic Floor Distress Inventory-20 (PFDI-20), Fear Avoidance Beliefs Questionnaire (Physical Activity/PA) and Female Sexual Function Index FSFI-19.

Feasibility of recruitment will be assessed by exploring: the number of those referred to the trial over the study period, who meet the eligibility criteria, the number of eligible patients who consent to participate in the trial over the study period,the number of patients who decline to participate, the number of participants who consent to participate that remain in the trial after 4-month follow-up, the number/proportion of participants with complete baseline data over the study period, the number/proportion of participants with complete follow-up data at 4 months follow-up, the number/proportion of participants retained at the end of each module of treatment.

Randomization Women with an injury in the levator found in the ultrasound will be randomized with a computer program into two groups, one for intervention and the other for control A group of women without injury will be invited to filling in the questionnaires that will be carried out in the study three, six months and one year postpartum.

Blinding Ultrasound diagnosis of levator ani muscle injury will be determined by 2 gynecologists blinded to delivery outcomes, using validated protocols. Women with levator ani injury will be randomly assigned to one of two groups: one (Intervention), and the other (the comparison group) receiving conventional recommendations.

The investigator assessing outcome will be blinded to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* simplex vaginal first delivery with a elevator ani injury
* aged ≥18 years
* understands the Swedish language in speech and writing
* approves vaginal examination

Exclusion Criteria:

* diagnosed sphincter injury grade 3-4
* serious postpartum disease (heart failure, thrombophlebitis, recent pulmonary embolism, acute infectious disease, genital haemorrhage, severe hypertension, dyspnoea, severe anemia or severe mental illness)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the trial. | 4 months after delivery
  The number of those referred to the trial over the study period, who meet the eligibility criteria, the number of eligible patients who consent to participate in the trial over the study period, and the number of patients who decline to participate, the number of participants who consent to participate that remain in the trial by 4-month follow-up, the number/proportion of participants with complete baseline data over the study period, the number/proportion of participants with complete follow-up data at 4 months follow-up, the number/proportion of participants retained at the end of each module of treatment.
Feasibility of the trial. | 6 months after delivery
  The number of those referred to the trial over the study period, who meet the eligibility criteria, the number of eligible patients who consent to participate in the trial over the study period, and the number of patients who decline to participate, the number of participants who consent to participate that remain in the trial by 4-month follow-up, the number/proportion of participants with complete baseline data over the study period, the number/proportion of participants with complete follow-up data at 4 months follow-up, the number/proportion of participants retained at the end of each module of treatment.
Feasibility of the trial. | 12 months after delivery
  The number of those referred to the trial over the study period, who meet the eligibility criteria, the number of eligible patients who consent to participate in the trial over the study period, and the number of patients who decline to participate, the number of participants who consent to participate that remain in the trial by 4-month follow-up, the number/proportion of participants with complete baseline data over the study period, the number/proportion of participants with complete follow-up data at 4 months follow-up, the number/proportion of participants retained at the end of each module of treatment.
Morphometry with ultrasound Area | 10-12 weeks after delivery
  3-D Ultrasound examination., Levator hiatus area at rest (cm2),during Valsalva (cm2) and at maximum contraction (cm2)
Morphometry with ultrasound Area | 12 months after delivery
  3-D Ultrasound examination., Levator hiatus area at rest (cm2),during Valsalva (cm2) and at maximum contraction (cm2)
Morphometry with ultrasound Levator urethra GAP (LUG) | 10-12 weeks after delivery
  The distance between the center of the urethra and the levator insertion (LUG) in cm
Morphometry with ultrasound Levator urethra GAP (LUG) | 12 months after delivery
  The distance between the center of the urethra and the levator insertion (LUG) in cm
Morphometry with ultrasound muscle thickness | 10-12 weeks after delivery
  Right and left puborectal muscle thickness (mm) .
Morphometry with ultrasound muscle thickness | 12 months after delivery
  Right and left puborectal muscle thickness (mm) .
Urogynecological symptoms. | 3 months after delivery
  Pelvic Floor Impact Questionnaire (PFIQ-7)
Urogynecological symptoms. | 6 months after delivery
  Pelvic Floor Impact Questionnaire (PFIQ-7)
Urogynecological symptoms. | 12 months after delivery
  Pelvic Floor Impact Questionnaire (PFIQ-7)
Urogynecological symptoms. | 3 months after delivery
  Pelvic Floor Distress Inventory-20 (PFDI-20)
Urogynecological symptoms. | 6 months after delivery
  Pelvic Floor Distress Inventory-20 (PFDI-20)
Urogynecological symptoms. | 12 months after delivery
  Pelvic Floor Distress Inventory-20 (PFDI-20)
Physics activity level. | 3 months after delivery
  Open questions on Physics activity level.
Physics activity level. | 6 months after delivery
  Open questions on Physics activity level.
Physics activity level. | 12 months after delivery
  Open questions on Physics activity level.
Sexual Function. | 3 months after delivery
  Female Sexual Function Index FSFI-19 questionnaire
Sexual Function. | 6 months after delivery
  Female Sexual Function Index FSFI-19 questionnaire
Sexual Function. | 12 months after delivery
  Female Sexual Function Index FSFI-19 questionnaire
Fear Avoidance Beliefs Questionnaire (Physical Activity/PA) | 3 months after delivery
  Fear-Avoidance Beliefs Questionnaire
Fear Avoidance Beliefs Questionnaire (Physical Activity/PA) | 6 months after delivery
  Fear-Avoidance Beliefs Questionnaire
Fear Avoidance Beliefs Questionnaire (Physical Activity/PA) | 12 months after delivery
  Fear-Avoidance Beliefs Questionnaire

SECONDARY OUTCOMES:
Pelvic Organ Prolapse Quantification Examination (POP-Q) | 10-12 weeks after delivery
  assessing the degree of prolapse of pelvic organs to help standardize diagnosing, comparing, documenting, and sharing of clinical findingsThe prolapsed organs will be measured in centimeters to the hymen
Pelvic Organ Prolapse Quantification Examination (POP-Q) | 12 months after delivery
  assessing the degree of prolapse of pelvic organs to help standardize diagnosing, comparing, documenting, and sharing of clinical findingsThe prolapsed organs will be measured in centimeters to the hymen
Age | 10-12 weeks after delivery
  Age in years
Body mass index (BMI) | 10-12 weeks after delivery
  BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2
Body mass index (BMI) | 12 months after delivery
  BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2
Weight gain during pregnancy | 10-12 weeks after delivery
  Weight gain during pregnancy in kilograms
Delivery mode | 10-12 weeks after delivery
  Delivery mode:vaginal delivery, forceps delivery or vacuum delivery
Baby's birth weight | 10-12 weeks after delivery
  Baby's birth weight in kilograms
Previous abdominal operation | 10-12 weeks after delivery
  Number of previous abdominal operation
Gastric bypass | 10-12 weeks after delivery
  Gastric bypass surgery
Modified Oxford Grading Scale | 10-12 weeks after delivery
  The modified Oxford Grading Scale [4] quantifies pelvic floor muscle strength as: 0, no contraction; 1, flicker; 2, weak; 3, moderate; 4, good; and 5, strong.
Modified Oxford Grading Scale | 6 months after delivery
  The modified Oxford Grading Scale [4] quantifies pelvic floor muscle strength as: 0, no contraction; 1, flicker; 2, weak; 3, moderate; 4, good; and 5, strong.
Modified Oxford Grading Scale | 12 months after delivery
  The modified Oxford Grading Scale [4] quantifies pelvic floor muscle strength as: 0, no contraction; 1, flicker; 2, weak; 3, moderate; 4, good; and 5, strong.

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Montejo, PhD, Principal Investigator — Vastra Gotaland Region
Locations (1):
- Nu sjukvård, Trollhättan, Sweden

IPD SHARING:
Plan to Share IPD: No